CLINICAL TRIAL: NCT07048119
Title: Development, Usability and Feasibility Pilot Study of a Videogame Aiming to Stimulate Cognitive and Non-cognitive Skills Among Low-income Preschoolers in Chile
Brief Title: Development, Usability and Feasibility Pilot Study of a Videogame
Acronym: Japi-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de los Andes, Chile (Other)
Collaborators: King's College London (Other); University of Talca (Other)
Responsible Party: Principal Investigator, Jorge Gaete, Full Professor, Universidad de los Andes, Chile
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UAN 201701
Record Dates: First submitted 2025-02-26; First posted 2025-07-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Mental Health Issue; Development, Child; Cognitive Ability, General
Keywords: Cognitive skills; Non-cognitive skills; Mental health; Preschoolers; Video game
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Intervention versus Treatment as Usual
Who Masked: Outcomes Assessor
Masking Description: Statistician was blinded to the group allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Japi 1.0 Intervention (Experimental): Video game of 10 sessions with activities stimulating cognitive (working memory and inhibitory control) and non-cognitve (emotion recognition and social competence) skills. Children will play with the game two times a week, each lasting 30 minutes, over 5 weeks. Sessions numbers 1 to 5 were focused on emotional recognition and inhibitory control. Sessions numbers 6 to 10 worked on working memory and social competence. Each session had eight activities and five tasks per activity with increasing difficulty levels.
  Interventions: Behavioral: Japi 1.0
- Control (No Intervention): The control group receives standard school curricula.

INTERVENTIONS:
Behavioral: Japi 1.0 — The intervention has ten sessions, and two sessions of 30 minutes were delivered each week for 5 weeks. Sessions numbers 1 to 5 were focused on emotional recognition and inhibitory control. Sessions numbers 6 to 10 worked on working memory and social competence. Each session had eight activities and five tasks per activity with increasing difficulty levels.
  Arms: Japi 1.0 Intervention

SUMMARY:
Mental health disorders are one of the leading causes of illness globally. The importance of psychosocial skills acquired in early childhood, such as executive functions, inhibitory control, emotional regulation, and social problem-solving, in preventing mental disorders has been reported. Furthermore, mental health care delivery is evolving, and mobile technology is becoming the medium for assessment and intervention. We developed Japi 1.0, a video game, to stimulate cognitive and non-cognitive skills in early childhood. This study aims to assess the functionality of this video game, student engagement and behavior, classroom climate, the feasibility of the implementation of the study and to explore the impact of the video game on the development of cognitive and non-cognitive skills.

DETAILED DESCRIPTION:
The use of technology in preventive interventions allows, on the one hand, the development of cost-effective strategies and, on the other, access to a large population. There are a number of therapeutic and preventive initiatives that have begun to be used in the mental health field in adolescents and adults. These interventions have been delivered through websites or mobile applications, and have shown some effectiveness. However, there are no studies on using these technologies in preschool populations. There is consensus in the scientific community that the stimulation of cognitive and non-cognitive skills in the first years of life promotes development in general and produces a beneficial impact in the long term on health and on different economic indicators.

The objectives of this research are: 1) To develop a video game prototype to be used on tablets by pre-kindergarten students from socio-economically vulnerable schools, which allows stimulating working memory, behavioral inhibition, emotion recognition, and social problem-solving skills in such a way as to prevent the development of behavioral problems and general psychological distress; 2) To carry out a pilot cluster Randomized Controlled Trial to evaluate several aspects of functionality of this video game, student engagement and behavior, classroom climate, the feasibility of the implementation of the study and to explore the impact of the video game on the development of cognitive and non-cognitive skills.

It is expected to recruit eight schools with at least one pre-kindergarten class, with an average of 30 students per class. Schools will be randomly allocated to intervention and control groups in a ratio of 1:1. The control group will receive their usual curricular activities. Meanwhile, the students in the intervention group will play the ten 30-minute video game sessions supervised by preschool teachers and research assistants. The frequency of sessions is expected to be twice a week for 5 weeks. Both groups will be evaluated at the beginning and after implementing Japi 1.0. The assessment will include the direct in-person measurement of working memory, behavioral inhibition, emotion recognition, and social problem-solving skills among children and evaluating children's emotional and behavioral problems rated by parents or caregivers. As the primary outcomes of this study are the evaluation of the functionality of this video game, student engagement, and behavior during playing, classroom climate, and the feasibility of the implementation of the study, the research team has developed quantitative and qualitative measures to collect this data.

ELIGIBILITY:
Inclusion Criteria Schools:

* Schools located in Santiago (Chile).
* Schools with Preschool Education.
* Mixed-sex schools.
* Schools with high vulnerability (≥ 75%), as stated in the School Vulnerability Index - National System of Equality Allocation (IVE-SINAE). This index is the proportion of high-vulnerability students in a given school, considering socioeconomic variables such as the mother's educational level, the father's educational level, and total monthly household income, among others.

Exclusion Criteria Schools:

* Four or more classes in Preschool. This criterion was considered for economic and practical reasons.
* Implementing a manualized program to promote cognitive or social-emotional skills.
* Participating in a similar study.

Inclusion Criteria for Students:

- Children attending pre-kindergarten (aged around 4 years old).

Exclusion criteria for Students

* Children with intellectual disability.
* Children unable to understand and speak Spanish

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 317 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-12-15 (Actual); Study Completion 2018-12-15 (Actual)

PRIMARY OUTCOMES:
Functionality of video game: Mechanical errors | Through study completion, an average of 1 year
  The number of errors in the video game (e.g., wrong interface, stuck or frozen screen, wrong reward stimulus after students´ correct responses) registered for tasks and activities during sessions.
Functionality of video game: Failure to record data in the server | Through study completion, an average of 1 year
  The number of students whose data from video game play was not recorded in the server.
Poor student engagement | Through study completion, an average of 1 year
  Percentage of students who lack attention and engagement and prematurely stop playing, making them unable to finish the tasks and activities during each session.
Feasibility: number of eligible schools | Through study completion, an average of 1 year
  The number of eligible schools, those contacted, and those who agreed to participate.
Feasibility: Participant recruitment | Through study completion, an average of 1 year
  The number of parents/caregivers and students who were contacted and those who consented and agreed to participate.
Feasibility: Attrition | Through study completion, an average of 1 year
  The number of participants' losses during the study.
Feasibility: Intervention duration | Through study completion, an average of 1 year
  Data will be collected on the time needed to complete the intervention.
Feasibility: Time requirement needed for measurements | Through study completion, an average of 1 year
  Time invested in baseline and after-intervention measurements.
Feasibility: Student attandance | Through study completion, an average of 1 year
  We will collect student attendance data by session to play with Japi 1.0.

SECONDARY OUTCOMES:
Working Memory: Corsi Block Test | Through study completion, an average of 1 year
  This test assesses visuospatial short-term working memory. It involves repeating a sequence of up to nine identical spatially separated blocks on a screen. The sequence starts simple but becomes more complex until the subject's performance declines. This number is known as the Corsi Span. The higher the score, the better the skill.
Working Memory: Woodcock- Muñoz Auditive Working Memory test | Through study completion, an average of 1 year
  A sequence of audio messages of words and numbers of increased difficulty is presented, and the child is requested to remember these sequences-the higher the score, the better the skill.
Inhibitory control: The Hearts and Flowers task | Through study completion, an average of 1 year
  The Hearts and Flowers task combines elements of Simon and spatial Stroop tasks. Children must follow the rule for congruent trials: "Press on the same side as the stimulus (Hearts)." For incongruent trials, children must follow the rule: "Press on the side opposite the stimulus (Flowers)." It requires working memory and inhibition control. The higher the score, the better the skill.
Executive function: The Minnesota Executive Function Scale (MEFS) | Through study completion, an average of 1 year
  This instrument evaluates executive functions, specifically cognitive flexibility, working memory, and inhibitory control, among individuals beginning at 24 months and extending throughout their lifespan. It is an adaptive virtual card-sorting task delivered on a tablet (4-minute average test duration). The higher the score, the better the skill.
Emotion recognition: Assessment of Children's Emotions Skills (ACES) | Through study completion, an average of 1 year
  It consists of a facial expressions task aiming to evaluate emotion expression knowledge and whether the subjects exhibit any anger bias. The 26-item scale consists of color photographs of ethnically diverse elementary schoolchildren depicting four expressions of the four basic emotions (happy, sad, angry, and scared) and 10 images of children without obvious facial expressions. The examiner shows the child the photographs one at a time and each time asks, "Is the child in the picture happy, sad, angry, or scared?" Then, the examiner registers the child's answer. The emotion accuracy score reflects how many items the children answer correctly (16 points is the perfect score). The higher the score, the better the skill. Additionally, there is an anger bias score, which is the number of times the children incorrectly identify the faces as displaying anger. The higher the score, the higher the anger bias.
Social competence: Challenging Situations Task (CST) | Through study completion, an average of 1 year
  This instrument evaluates the ability of children to solve social problems. The children are presented with six vignettes that describe problems between peers. Following the presentation of each challenging situation, four pictures of happy, sad, angry, and neutral affect are presented in random order. The child is asked to point to the picture that best describes how they feel when [one of the situations] happens. Then, four pictures of behavioral responses (prosocial, aggressive, disruptive, or less adaptative behavior [cry], and avoidant) are presented in random order, and the child is asked, "What do you do in this situation]?" The answers are categorized into four possibilities: prosocial, aggressive, cry, and avoidant. Scores for affective and behavioral responses used are the number of times each affect, and each behavioral response is chosen by each child across the six situations. The higher the prosocial behavioral response score, the better the skill.
Behavioral problems and psychological assessment: The Strengths and Difficulties Questionnaire (SDQ). | Through study completion, an average of 1 year
  This 25-question questionnaire explores different symptoms grouped into 5 sub-scales (with 5 items each): (1) emotional symptoms, (2) behavioral problems, (3) problems with peers, (4) symptoms of lack of attention and hyperactivity, and (5) prosocial skills. The first four sub-scales refer to children's difficulties and may be grouped into a general sub-scale of difficulties (20 items). The sub-scale of prosocial skills refers to positive and adaptive behaviors in relationships. Each item is answered on a scale of responses from 1=not true to 3=absolutely true. There is a version for Educators and parents (to evaluate children from 4 to 16 years old) and a self-report for teenagers (ages 11 to 16 years old). The Parents' version of this instrument will be used-the higher the score in the total difficulties sub-scale, the higher the behavior problems in the case of the prosocial sub-scale; the higher the score, the higher the prosocial skill.

CONTACTS AND LOCATIONS:
Overall Officials: Jorge E Gaete, MD. PhD., Study Director — Universidad de Los Andes
Locations (1):
- Universidad de los Andes, Santiago, Las Condes, Chile

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to ethical considerations, however tha data as a whole will be available on request to the Principal Investigator.

REFERENCES:
- [Background] Carlson S, Zelazo P. Minnesota executive function scale: Test manual. Saint Paul, MN: Reflection Sciences. 2014.
- [Background] Goodman R. Psychometric properties of the strengths and difficulties questionnaire. J Am Acad Child Adolesc Psychiatry. 2001 Nov;40(11):1337-45. doi: 10.1097/00004583-200111000-00015. PMID 11699809
- [Background] Goodman R. The Strengths and Difficulties Questionnaire: a research note. J Child Psychol Psychiatry. 1997 Jul;38(5):581-6. doi: 10.1111/j.1469-7610.1997.tb01545.x. PMID 9255702
- [Background] Denham SA, Way E, Kalb SC, Warren-Khot HK, Bassett HH. Preschoolers' social information processing and early school success: the challenging situations task. Br J Dev Psychol. 2013 Jun;31(Pt 2):180-97. doi: 10.1111/j.2044-835X.2012.02085.x. Epub 2012 Sep 27. PMID 23659890
- [Background] Chung C, Choi S, Bae J, Jeong H, Lee J, Lee H. Developing and Validating a Korean Version of the Assessment of Children's Emotional Skills. Child Psychiatry Hum Dev. 2024 Jun;55(3):819-830. doi: 10.1007/s10578-022-01452-2. Epub 2022 Oct 13. PMID 36229629
- [Background] Davidson MC, Amso D, Anderson LC, Diamond A. Development of cognitive control and executive functions from 4 to 13 years: evidence from manipulations of memory, inhibition, and task switching. Neuropsychologia. 2006;44(11):2037-78. doi: 10.1016/j.neuropsychologia.2006.02.006. Epub 2006 Mar 31. PMID 16580701
- [Background] Gathercole SE, Willis CS, Baddeley AD, Emslie H. The Children's Test of Nonword Repetition: a test of phonological working memory. Memory. 1994 Jun;2(2):103-27. doi: 10.1080/09658219408258940. PMID 7584287
- [Background] Orsini A. Corsi's block-tapping test: standardization and concurrent validity with WISC-R for children aged 11 to 16. Percept Mot Skills. 1994 Dec;79(3 Pt 2):1547-54. doi: 10.2466/pms.1994.79.3f.1547. PMID 7870543
- [Background] Doyle O, Harmon CP, Heckman JJ, Tremblay RE. Investing in early human development: timing and economic efficiency. Econ Hum Biol. 2009 Mar;7(1):1-6. doi: 10.1016/j.ehb.2009.01.002. Epub 2009 Jan 21. PMID 19213617
- [Background] Campbell F, Conti G, Heckman JJ, Moon SH, Pinto R, Pungello E, Pan Y. Early childhood investments substantially boost adult health. Science. 2014 Mar 28;343(6178):1478-85. doi: 10.1126/science.1248429. PMID 24675955
- [Background] Bucci S, Schwannauer M, Berry N. The digital revolution and its impact on mental health care. Psychol Psychother. 2019 Jun;92(2):277-297. doi: 10.1111/papt.12222. Epub 2019 Mar 28. PMID 30924316
- [Background] Garon N, Bryson SE, Smith IM. Executive function in preschoolers: a review using an integrative framework. Psychol Bull. 2008 Jan;134(1):31-60. doi: 10.1037/0033-2909.134.1.31. PMID 18193994
- [Background] Berger A, Kofman O, Livneh U, Henik A. Multidisciplinary perspectives on attention and the development of self-regulation. Prog Neurobiol. 2007 Aug;82(5):256-86. doi: 10.1016/j.pneurobio.2007.06.004. Epub 2007 Jun 22. PMID 17651888
- [Background] Durlak JA, Weissberg RP, Dymnicki AB, Taylor RD, Schellinger KB. The impact of enhancing students' social and emotional learning: a meta-analysis of school-based universal interventions. Child Dev. 2011 Jan-Feb;82(1):405-32. doi: 10.1111/j.1467-8624.2010.01564.x. PMID 21291449
- [Background] Cunha F, Heckman J, Schennach S. Estimating the Technology of Cognitive and Noncognitive Skill Formation. Econometrica. 2010 May 1;78(3):883-931. doi: 10.3982/ECTA6551. PMID 20563300
- [Background] GBD 2019 Mental Disorders Collaborators. Global, regional, and national burden of 12 mental disorders in 204 countries and territories, 1990-2019: a systematic analysis for the Global Burden of Disease Study 2019. Lancet Psychiatry. 2022 Feb;9(2):137-150. doi: 10.1016/S2215-0366(21)00395-3. Epub 2022 Jan 10. PMID 35026139